CLINICAL TRIAL: NCT00368446
Title: Genetic Disorders of Mucociliary Clearance
Brief Title: Genetic Disorders of Mucociliary Clearance in Nontuberculous Mycobacterial Lung Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060217; 06-H-0217
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-07-08

CONDITIONS: Cystic Fibrosis; Pseudohypoaldosteronism; Nontuberculous Mycobacterial Infection; Chronic Granulomatous Disease; Primary Ciliary Dyskinesia
Keywords: Nontuberculous Mycobacterial Infection; Primary Ciliary Dyskinesia; Cystic Fibrosis; Pseudohypoaldosteronism; Chronic Granulomatous Disease; Natural History; Mycobacterial Infection; PCD; CF; PHA; Healthy Volunteer; HV
MeSH Terms: conditions — Cystic Fibrosis; Pseudohypoaldosteronism; Granulomatous Disease, Chronic; Ciliary Motility Disorders; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Normal
- 2: patients with Genetic Disorders of Mucociliary Clearance

SUMMARY:
Healthy volunteers and patients with diseases that involve problems clearing mucus from the lungs will be examined and tested to better understand the reasons for recurring lung infections in these patients and to try to develop better ways to diagnose and treat them. The study will also try to identify the genes responsible for these diseases.

Healthy volunteers 18 years of age and older and patients 2 years of age or older with suspected primary ciliary dyskinesia (PCD), variant cystic fibrosis (CF) or pseudohypoaldosteronism (PHA) may be eligible for this study. Patients enrolled in the Natural History Study of Nontuberculous Mycobacteria at NIH or other NIH natural history protocols may also be enrolled. Participants undergo the following tests and procedures during a 1-day visit at the NIH Clinical Center, as follows:

All patients and normal volunteers have the following procedures:

* Physical examination and review of medical and genetic history and family genetic history.
* Lung function test and measurement of oxygen saturation level.
* Nitric oxide measurement to measure the amount of nitric oxide production in the nose: A small tube is placed in the nose while the subject breathes through the mouth into a cardboard tube.

All patients have the following additional procedures:

* Blood tests for liver and kidney function, blood count, immunoglobulins and pregnancy test (where appropriate).
* Blood test or buccal scrape (brushing the inside of the cheek) to obtain DNA to look for gene mutations that cause PCD, CF or PHA.
* Scrape biopsy of cell lining the inside of the nose: A small toothpick-sized plastic stick with a tiny cup on the end is used to get nasal lining cells to look at the cilia (hair-like structures that move mucus).
* Semen analysis (in some men) to test sperm tail function or structure.

Patients suspected of having a variant of CF or PHA, including nontuberculous mycobacterial lung disease, have the following additional procedures:

* Sweat chloride test: A medicine is placed on the arm to produce sweat; then, a very low level of electric current is applied for 5 to 12 minutes. Sweat is collected in a plastic tube and tested for salt content.
* Blood draw for CF genetic testing, if necessary, and to measure levels of the enzyme trypsin.
* Saliva collection to measure sodium and chloride content.
* Nasal potential difference to measure the electrical activity of the cells lining the inside of the nose: A soft plastic tube filled with a salt solution is passed into the nasal passage and a sterile needle is placed under the skin of the arm. This test provides information about how the lining of the nose is able to get used to changes in temperature and humidity. (Normal volunteers also have this test.)

DETAILED DESCRIPTION:
Background: Nontuberculous mycobacteria (NTM) are ubiquitous environmental organisms that have been increasingly associated with human disease, commonly involving the lung. Post menopausal Caucasian women seem particularly predisposed to the development of peripheral nodules and dilated airways (bronchiectasis) associated with these organisms. These women have distinguishing body characteristics of being taller and thinner than age and gender matched controls yet have no identifiable systemic immune defects. There is, however, considerable overlap with genetic disorders of mucociliary clearance such as cystic fibrosis (CF) and primary ciliary dyskinesia (PCD). The Genetic Diseases of Mucociliary Clearance Consortium (GDMCC) is one of 10 consortia in the Rare Diseases Clinical Research Network formed under the Office of Rare Diseases in collaboration with NCRR, NICHD, NINDS, NIAMS, NIDDK, NHLBI in response to the Rare Diseases Act of 2002. The GDMCC is comprised of 5 geographically-dispersed clinical research sites that are designed to study rare diseases which involve defects in clearance of mucus secretions from the airways (defective "mucociliary clearance"). These sites will collaborate in diagnostic, genetic, and other studies in patients with impairments of mucociliary clearance, including primary ciliary dyskinesia (PCD), variant cystic fibrosis (CF), and pseudohypoaldosteronism (PHA). These studies are also applicable to diseases where altered airways clearance may play a primary or contributory role such as nontuberculous mycobacterial lung disease, chronic granulomatous disease, and the hyper-IgE syndromes. Disorders such as PCD, CF, and PHA reflect genetic defects in airway host-defense, and typically result in chronic infection of the airways. Patients with these disorders of the conducting airways and sinuses have delayed (or incorrect) diagnoses, because diagnostic tests are not readily available. These patients may also have sub-optimal management of their clinical disease, because the cause of these disorders is not well-defined, and treatment regimens are usually not driven by evidence-based medicine.

Aims: The major aim of this study is to employ a systematic approach to the diagnostic and functional evaluation of these patients with chronic airways disease in individual patients, better define host susceptibility to infections from environmental organisms such as the nontuberculous mycobacteria, and potentially lead to the development of better diagnostic techniques, including genetic testing. In addition, we will compare/contrast clinical features (phenotype) across these disorders. A rigorous cross-sectional comparison of the clinical features will provide better understanding of the clinical disease of these disorders; in turn this will lead not only to a better standard of clinical care, but will also assist in the identification of novel therapeutic approaches.

Methods: This is a cross-sectional diagnostic / mechanistic protocol to investigate airway host-defenses. The patient populations for these studies include individuals with recurring airway infections such as those with nontuberculous mycobacteria lung disease who may have defective airway host defenses as a predisposing factor, individuals carrying a tentative diagnosis of the three known genetic disorders of mucociliary clearance (PCD, variant CF, or PHA), and individuals suspected to have one of these disorders but with inadequate or inconclusive diagnostic tests. Individuals in this latter category must have a preliminary clinical evaluation to evaluate for other more common disorders that may have similar manifestations including classical CF, immunodeficiency, asthma, and severe gastroesophageal reflux. The evaluation will include a detailed assessment of clinical features; specialized laboratory measurements such as nasal potential difference to evaluate the function of chloride and sodium channels associated with CF and PHA, nasal biopsy specimens and nasal nitric oxide measurements to assess cilia structure and function which are abnormal in PCD; and genetic studies to identify disease - causing mutations in genes associated with CF, PCD, and PHA.

ELIGIBILITY:
* INCLUSION CRITERIA:

Overview: Inclusion criteria reflect the two-fold purpose of this protocol. It is primarily intended to evaluate the cohort of patients followed at the NIH Clinical Center under Protocol 01-I-0202, Natural History, Genetics, Phenotype, and Treatment of Mycobacterial Infections, and in this regard, the inclusion criteria mirror those of that protocol. Secondly it is part of the multicenter collaborative protocol as a participating site in the Genetic Disorders of Mucociliary Clearance Consortium, one of the Rare Disease Clinical Consortia sponsored by the Office of Rare Diseases. There is a clear-cut need for geographically dispersed centers to have expertise in the diagnostic evaluation and treatment of patients with rare diseases of the airways, including patients with suspected PCD, non-classical or variant CF, and PHA. The 5 sites will perform rigorous diagnostic evaluations utilizing innovative, but standardized methods (SOPs contained in Manual of Operations). As a participating site in the Consortium, we will cast a broad net to include as many participants as feasible. This will include a multi-center standardized diagnostic evaluation and clinical evaluation, giving us a better chance to define the clinical spectrum of disease.

The criteria for participants to enter this study mandates that each patient either be enrolled in the 01-I-0202, Natural History, Genetics, Phenotype, and Treatment of Mycobacterial Infections or related NIH Natural History Protocol, or if referred as part of the Consortium, have received a standard (current clinical practice) diagnostic evaluation that includes testing for asthma, severe gastroesophageal reflux and/or classic CF, prior to enrolling in the Consortium study. Healthy adult control participants will be enrolled for comparison assessment of noninvasive nasal nitric oxide and nasal potential difference measurements only. The health status of these control participants will be assessed with the standardized clinical history, family history, physical exam including height and weight, vital signs, oximetry, and spirometry measurements.

To enter the study, individuals with a suspected mucociliary clearance defect (n=100) must be age 2 years or older and meet one of the 4 following profiles:

1. Have known or suspected nontuberculous mycobacterial lung disease and enrolled in Protocol 01-I-0202, Natural History, Genetics, Phenotype, and Treatment of Mycobacterial Infections.
2. Have high suspicion for the diagnosis of PCD, based on ciliary ultrastructural changes on EM (if performed elsewhere prior to referral) or clinical features (chronic sinopulmonary disease, chronic otitis media, history of neonatal respiratory distress or situs inversus), or PCD in a sibling and one of the clinical features of PCD.
3. Have chronic sino-pulmonary disease with clinical features that overlap with variant CF and PCD, but with diagnostic tests to rule out classical CF (sweat Cl- testing and CF gene mutation screening). This may include patients with other known immune deficiencies such as chronic granulomatous disease followed on NIH natural history protocols.
4. Known or suspected PHA (or variant PHA), which might include elevated (or borderline) sweat Cl- values.

To enter the study as a healthy control (n=25), individuals must be age 18 or older and free of any known disease, chronic medical conditions, family history of cystic fibrosis or primary ciliary dyskinesia, or any cognitive impairment or significant disability that might preclude voluntary consent or the ability to safely comply with the instructions or sit through the testing.

EXCLUSION CRITERIA:

Persons who cannot be evaluated at the Clinical Center or who have severe cognitive impairment or other severe disability that precludes the ability to understand instructions or sit/lie still for the evaluation will be excluded. Certain conditions may preclude specific procedures included in the protocol, but may still allow pertinent parts of this diagnostic evaluation. These conditions/procedures may include: pregnancy/Chest PA/Lat x-ray; allergy to pilocarpine /sweat testing. For reversible conditions such as acute upper airway infection, significant epistaxis within the prior week (not related to #2 below), or lower airway infection with uncontrollable coughing, the participant may need to be rescheduled upon resolution.

For nasal nitric oxide and nasal potential difference measurements or nasal mucosal scrape biopsies:

1. Anatomic abnormality of the nose or sinuses (e.g. complete sinus blockage or turbinatectomy) that precludes either the measurement of nasal nitric oxide or nasal potential difference.
2. A severe bleeding diathesis or condition such as hereditary hemorrhagic telangiectasia syndrome that may predispose to significant nasal bleeding or result in severely excoriated nasal mucosa.
3. Inability to sit still for up to 15 minutes while the nasal catheters are held on the mucosal surface for transepithelial potential difference measurements. This would include the presence of acute or chronic lower respiratory tract infection that results in uncontrollable coughing.
4. Diffuse skin condition that would preclude placement of the subcutaneous reference electrode (butterfly needle) for nasal PD measurement.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are approximately 100 patients who have been referred to the Clinical Center at NIH, or who have contacted us directly for evaluation of nontuberculous mycobacterial lung disease. Most of these are post-menopausal Caucasian women. Some had known diagnoses of CF or PCD at the time of referral and others have been subsequently diagnosed with these disorders after evaluation here. This population likely reflects a concentrated source population of potential cases of PCD and variant CF to feed into the Consortium. Additionally, the Clinical Center will serve as a referral site for cases of suspected PCD, variant CF, and PHA who don't necessarily have nontuberculous mycobacterial infections. These referrals will likely be concentrated in the National Capital Area and constitute a minority of the patients evaluated on the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2006-10-17 (Actual)

PRIMARY OUTCOMES:
PCD compatible clinical phenotype or sibling with PCD, plus defect in ciliary ultrastructure | 6 years
  compatible clinical phenotype (sinopulmonary disease and/or neonatal respiratory disorder plus or minus situs inversus) or sibling with PCD, plus defect in ciliary ultrastructure (inner or outer dynein arm; radial spoke; central complex)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Lipton, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0217.html